CLINICAL TRIAL: NCT00637143
Title: Prograf® (Tacrolimus) as Secondary Intervention vs. Continuation of Cyclosporine in Patients at Risk for Chronic Renal Allograft Failure
Brief Title: Tacrolimus as Secondary Intervention vs. Continuation of Cyclosporine in Renal Transplant Patients With Chronic Renal Allograft Failure (CRAF)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Collaborators: Astellas Pharma Canada, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FKC-003
Record Dates: First submitted 2008-03-10; First posted 2008-03-17 (Estimated); Last update posted 2017-02-16 (Actual); Status verified 2017-02

CONDITIONS: Renal Transplantation; Chronic Renal Allograft Failure
Keywords: Renal transplant; Cyclosporine; Tacrolimus; Intervention; Interstitial Fibrosis Tubular Atrophy; Chronic Renal Allograft Failure
MeSH Terms: interventions — Tacrolimus; Cyclosporine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Oral
  Interventions: Drug: Tacrolimus
- 2 (Active Comparator): Oral
  Interventions: Drug: Cyclosporine

INTERVENTIONS:
Drug: Tacrolimus — Oral
  Other Names: FK506; Prograf
  Arms: 1
Drug: Cyclosporine — Oral
  Other Names: Neoral
  Arms: 2

SUMMARY:
The purpose of this study is to compare renal transplant recipients on cyclosporine maintenance therapy vs. those converted to tacrolimus-based immunosuppression with respect to renal outcomes.

DETAILED DESCRIPTION:
The objective of this study is to compare the incidence, progression and severity of chronic renal allograft failure in at-risk patients who are converted from cyclosporine to tacrolimus-based immunosuppression to patients who remain on cyclosporine.

ELIGIBILITY:
Inclusion Criteria:

* Patient is at least 3 months post-transplant of a cadaveric or living donor kidney
* Patient has been on a cyclosporine-based immunosuppression regimen since the transplant
* Patient has one of the following risk factors for chronic renal allograft failure at the baseline biopsy:

  * Serum creatinine: Male: >=2.0mg/dL (176.8 umol/L); Female: >= 1.7mg/dL (150.28 umol/L) 3 months or later post-transplant
  * Serum creatinine > 30% increased over post-discharge nadir
* Patient has had a renal biopsy > 3 months after transplant and within 6 months prior to enrollment
* Patient or legal guardian has signed and dated an IRB approved informed consent document
* Female patient has a negative pregnancy test and agrees to practice effective birth control while receiving mycophenolate mofetil (MMF)

Exclusion Criteria:

* Patient is dialysis dependent and has recurrence of primary or de novo renal disease
* Patient has an estimated creatinine clearance <25mL/min
* Patient has changed maintenance immunosuppressant therapy (e.g., azathioprine to MMF) within 3 months of randomization
* Baseline biopsy shows acute rejection Grade >=IIB using Banff 95 criteria or >= Grade IIA using Banff 97 criteria
* Patient requires antilymphocyte therapy to treat rejection at baseline or post-baseline biopsy
* Patient has received an investigational immunosuppressant within 3 months, or has a known hypersensitivity to tacrolimus, or any excipients of the drug
* Patient is a known carrier of any of the HIV viruses

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 1999-04; Primary Completion 2006-02 (Actual); Study Completion 2006-02 (Actual)

PRIMARY OUTCOMES:
Graft Survival | 5 years

SECONDARY OUTCOMES:
Patient Survival | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Central Contact, Study Chair — Astellas Pharma Canada, Inc.
Locations (11):
- Canada (11):
  - Calgary, Alberta
  - Edmonton, Alberta
  - Vancouver, British Columbia
  - Winnipeg, Manitoba
  - St. John's, Newfoundland and Labrador
  - Halifax, Nova Scotia
  - Hamilton, Ontario
  - London, Ontario
  - Toronto, Ontario
  - Montreal, Quebec
  - Saskatoon, Saskatchewan

REFERENCES:
- [Background] Jevnikar A, Arlen D, Barrett B, Boucher A, Cardella C, Cockfield SM, Rush D, Paraskevas S, Shapiro J, Shoker A, Yilmaz S, Zaltzman JS, Kiberd B. Five-year study of tacrolimus as secondary intervention versus continuation of cyclosporine in renal transplant patients at risk for chronic renal allograft failure. Transplantation. 2008 Oct 15;86(7):953-60. doi: 10.1097/TP.0b013e318186dd0c. PMID 18852662
- See also: Link to results on Astellas Clinical Study Results website — https://www.astellasclinicalstudyresults.com/study.aspx?ID=154